CLINICAL TRIAL: NCT06923410
Title: Multilingual Exploration of the Clinical Intelligent Management System Based on a Multimodal Foundation Model
Brief Title: Clinical Intelligent Management System - Multilingual Exploration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tsinghua University (Other)
Responsible Party: Principal Investigator, Tien Yin Wong, Professor, Tsinghua University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24694-4-01
Record Dates: First submitted 2025-04-02; First posted 2025-04-11 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Primary Care Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI Agent Doctor group (Active Comparator): Standardized simulated patients consult with AI Agent Doctor, providing AI-generated diagnoses and treatments for health care.
  Interventions: Device: AI model
- Primary care physicians groups (No Intervention): Standardized simulated patients consult with physicians, providing routine diagnoses and treatments as their usual standard health care.

INTERVENTIONS:
Device: AI model — The clinical intelligent AI system is equipped with an AI agent doctor, enabling patients to conduct self-consultations and receive care anytime and anywhere without the need for a real doctor.
  Arms: AI Agent Doctor group

SUMMARY:
This study aims to explore the diagnostic and therapeutic performance of a multimodal foundation model-based clinical intelligent management system in simulated outpatient scenarios. Specifically, it will compare the system's AI agent with general practitioners from different linguistic and cultural backgrounds worldwide, as well as various dialect and minority language regions in China.

The study will be conducted across multiple centers in diverse regions to comprehensively evaluate the system's adaptability. Using a prospective, single-blind design, each center will recruit primary care physicians.

Standardized simulated patients across all centers will be trained based on the same set of standardized cases and then will consult with four real physicians and the AI agent, ensuring consistency.

By comparing diagnostic and treatment quality, patient satisfaction, and clinical outcomes, this study aims to explore the system's effectiveness in enhancing primary care and patient management across different regions and linguistic environments.

ELIGIBILITY:
Inclusion criteria for primary care physicians:

* Fluent in the local languages spoken at each center.
* With the general practice medical qualifications.
* Agree to participate in the study and sign the informed consent form.

Inclusion criteria for simulated patient volunteers:

* Age ≥ 18 years.
* Fluent in the local languages spoken at each center.
* Able to use electronic devices with intelligent systems.
* Able to accurately express symptoms and participate throughout the process.
* Agree to participate in the study and sign the informed consent form.

Exclision criteria: N/A

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Assessment of physician's clinical abilities | Immediately after the simulated consultation
  Clinical Abilities Assessment Scales for Primary Care (range: 0 to 100 for each case; the higher scores means the better performance)

SECONDARY OUTCOMES:
System's Usability | Immediately after the simulated consultation with AI system
  System Usability Evaluation Scale accessed by participating simulated patients, rated on a five-point Likert scale from strongly disagree (1) to strongly agree (5). (A higher scale value indicates higher perceived usability of the technology.)

CONTACTS AND LOCATIONS:
Locations (1):
- Tiantongyuan North Community Healthcare Center, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No